CLINICAL TRIAL: NCT03264404
Title: Phase II Open-Label, Single-Center Study Evaluating Safety and Efficacy of Pembrolizumab Following Induction With the Hypomethylating Agent Azacitidine in Patients With Advanced Pancreatic Cancer After Failure of First-Line Therapy
Brief Title: Azacitidine and Pembrolizumab in Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Susan E. Bates (Other)
Responsible Party: Sponsor-Investigator, Susan E. Bates, Professor of Medicine and Assistant Attending in Hematology / Oncology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR3554
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Results first posted 2023-07-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pancreas Cancer
Keywords: Pancreas; pembrolizumab; azacitidine; metastatic pancreatic cancer; first-line
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pembrolizumab; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab (Experimental): Patients with advanced pancreatic cancer will receive pembrolizumab with the hypomethylating agent azacitidine.
  Interventions: Drug: Pembrolizumab; Drug: Azacitidine

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV every 3 weeks until progression
  Other Names: Keytruda
Drug: Azacitidine — 50 mg/m2 subcutaneous daily for 5 days every 28 days
  Other Names: Vidaza

SUMMARY:
The purpose of this study is to determine the effectiveness of combining immune therapy, pembrolizumab, with a hypomethylating agent, azacitidine, for pancreatic cancer. People who have advanced pancreatic cancer with disease progression on first-line therapy are usually treated with a second chemotherapy regimen. However, there is no single accepted chemotherapy regimen and national guidelines recommend chemotherapy or clinical trial participation. In this study, all study subjects will receive a combination of immune therapy (every 3 weeks) and a hypomethylating agent (every 4 weeks). To date, studies have shown that combining a hypomethylating agent with chemotherapy or immune therapy may benefit patients across different solid tumor types including pancreatic cancer. Preclinical data in a mouse model of pancreatic cancer demonstrates improvement in survival with the combination of a hypomethylating agent and immune therapy. However, the use of single agent hypomethylating agent or immune therapy has not been shown to be effective in patients with pancreatic cancer. The one exception, to date, is the use of immune therapy in those individuals with a particular genetic feature known as mismatch repair deficiency and microsatellite instability. The combination of immune therapy and a hypomethylating agent has not been studied in human subjects and is not approved by the FDA for use in pancreatic cancer.

This is a non-randomized, single-center, open-label trial of pembrolizumab and azacitidine in subjects with locally advanced or metastatic pancreatic adenocarcinoma. Approximately 31 individuals will be asked to participate in this study.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDA) has the worst prognosis of any major malignancy in the United States and, unlike other common cancers, annual deaths from PDA are rising. Despite recent advances, cytotoxic chemotherapy for PDA has been disappointing. Even among the small subset of patients who are suitable for surgical resection at the time of diagnosis, complete resection is followed by recurrence in majority of patients without further systemic therapy. Thus all PDA patients require systemic chemotherapy and more effective regimens are urgently needed.

Combination chemotherapy is effective in controlling disease and prolonging survival in patients with advanced pancreatic cancer. Despite recent successful phase 3 studies in the first-line setting, there is no defined second-line treatment for patients who experience disease progression following first-line therapy. Consensus guidelines (such as the National Comprehensive Cancer Network (NCCN) guidelines) recommend clinical trial participation in this setting.

The investigators' pre-clinical data suggests that decitabine treatment in the KPC model of pancreatic cancer leads to a significant up-regulation of interferon-related genes and a polarization of the infiltrating immune cells. Based on these results, the investigators have evaluated the effect of single agent decitabine or anti-PD1H (a homologue of PD1 with very similar function and expression pattern) compared to combination therapy (treatment with decitabine followed by PD1H blockade). The investigators' preliminary results showed minimal effect of either agent alone on tumor growth but marked decrease in tumor progression in the combination arm. These results form the foundation of this phase II study.

This study will treat patients with the combination of azacitidine and pembrolizumab. A direct comparison between azacitidine and decitabine in terms of efficacy within a controlled clinical trial has not been performed thus far. In randomized myelodysplastic syndrome (MDS) trials, the remission rates were similar for azacitidine and decitabine but the overall survival in the experimental arm was significantly shorter in the decitabine trial compared to the azacitidine trial. A primary reason to utilize azacitidine in this setting is our desire to amply reduced dose therapy with the goal of maintaining subjects on therapy Low-dose azacitidine is being tested in phase I/II clinical trials for advanced solid tumors-mainly colorectal cancer, small-cell lung carcinomas, ovarian cancer, and breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Age ≥18 years of age on day of signing informed consent.
* Have confirmed diagnosis of pancreatic ductal adenocarcinoma
* Have a predicted life expectancy of greater than 3 months.
* Have measurable disease based on RECIST 1.1.
* Have a performance status of 0 or 1 using the Eastern Cooperative Oncology Group (ECOG) Performance Scale within 3 days of first dose of study drug.
* Have documented radiographic progression to or documented intolerance of first line systemic chemotherapy which included either gemcitabine or Fluorouracil (5-FU) based regimen (including capecitabine).
* Subjects who have documented disease recurrence within 6 months of completing neoadjuvant or adjuvant chemotherapy for limited disease will be eligible for study. Subjects who recur greater than 6 months after completing adjuvant or neoadjuvant chemotherapy will not be eligible unless they receive additional chemotherapy for advanced disease.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy, or herbal/complementary oral or IV medicine within 2 weeks of the first dose of treatment.
* Has received chemotherapy or radiotherapy within 14 days of first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Bates, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 36
Completed | 2
Not Completed | 34
Not completed — Death | 2
Not completed — Physician Decision | 1
Not completed — Disease Progression | 28
Not completed — Adverse Event | 1
Not completed — Off study prior to treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 28
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the first day of trial treatment to the first documented disease progression per RECIST 1.1 (At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression)) or death due to any cause, whichever occurs first.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 36
months | 1.49 [1.38 to 1.74]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of the participants in the analysis population who have a complete response (CR) or partial response (PR). Responses are based on assessments per RECIST 1.1.
Time Frame: Throughout study duration, up to approx 80 months
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 31
percentage of participants | 9.7

3. Secondary Outcome: Duration of Response (DOR)
Description: For subjects who demonstrate CR or PR, based on assessments per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Time Frame: Throughout study duration, up to approx 80 months
Population: 3 participants had a complete or partial response to treatment, so this outcome measure was assessed in those 3 patients only.
Measure: Number; unit: days
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 3
days
  Patient 1 | 2274
  Patient 2 | 881
  Patient 3 | 28

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants who have achieved CR, PR, or stable disease (SD) based on assessments per RECIST 1.1.
Time Frame: Throughout study duration, up to approx 80 months
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 31
percentage of participants | 35.5

ADVERSE EVENTS:
Time Frame: Throughout study duration, up to approx 80 months
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 26/36
Serious Adverse Events (participants affected / at risk) | 9/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=36)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Gastric hemorrhage (General disorders) | 2 (2)
Endocrine disorders (Endocrine disorders) | 1 (2)
Nervous system disorders (Nervous system disorders) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Vascular disorders (Vascular disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (4)
Ascites (Gastrointestinal disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Thromboembolic event (Vascular disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=36)
Vomiting (Gastrointestinal disorders) | 5 (7)
Abdominal Pain (Gastrointestinal disorders) | 9 (13)
Diarrhea (Gastrointestinal disorders) | 13 (21)
Alanine aminotransferase increase (Investigations) | 5 (9)
International Normalized Ratio (INR) Increased (Investigations) | 1 (3)
Hyponatremia (Investigations) | 5 (6)
Hypercalcemia (Investigations) | 1 (1)
Creatinine Increased (Investigations) | 1 (2)
Hyperkalemia (Investigations) | 3 (4)
Hypoalbuminemia (Investigations) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Alkaline phosphatase increased (Investigations) | 7 (17)
Pain (General disorders) | 3 (3)
Chills (General disorders) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 5 (10)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 7 (12)
Bloating (Gastrointestinal disorders) | 7 (11)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)
Hepatobiliary disorder (Hepatobiliary disorders) | 1 (2)
Cough (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 2 (2)
Fatigue (General disorders) | 8 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Constipation (Gastrointestinal disorders) | 12 (13)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Injection site reaction (General disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 6 (7)
Anorexia (Metabolism and nutrition disorders) | 9 (13)
Hypokalemia (Investigations) | 3 (9)
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 4 (10)
Fever (General disorders) | 2 (2)
Chest wall pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Platelet count decreased (Investigations) | 2 (4)
Infections and infestations (Infections and infestations) | 6 (8)
Acute kidney injury (Renal and urinary disorders) | 2 (3)
Weight loss (Investigations) | 4 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Sore throat (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Hypothyroidism (Endocrine disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (3)
Confusion (General disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (4)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (8)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Portal hypertension (Hepatobiliary disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Hypernatremia (Investigations) | 1 (1)
Endocrine disorders (Endocrine disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Sepsis (Infections and infestations) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Edema, Limbs (General disorders) | 2 (2)
Hot flashes (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Stroke (Nervous system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Hypocalcemia (Investigations) | 1 (1)
Hypomagnesemia (Investigations) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Cardiac troponin T increased (Investigations) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Weight gain (Investigations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT03264404/Prot_SAP_001.pdf